CLINICAL TRIAL: NCT05510050
Title: Comparison Study of Manapol and DaltonMax on Immune Function, Microbiome, and Related Variables in Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Collaborators: Mannatech (Unknown)
Responsible Party: Principal Investigator, Richard Bloomer, Dean of the College of Health Sciences, University of Memphis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PRO-FY2022-131
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Microbiome; Immune Function
Keywords: Aloe Vera extract; Manapol; Dalton Max

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo controlled
Who Masked: Participant, Investigator
Masking Description: Conditions will be provided in blinded containers (e.g. A,B,C).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Manapol (Experimental): 1000 mg (Manapol only) Aloe Vera extract daily
  Interventions: Dietary Supplement: Aloe Vera Extract 1
- Dalton Max (Experimental): 1000 mg (Dalton Max only) Aloe Vera extract daily
  Interventions: Dietary Supplement: Aloe Vera Extract 2
- Placebo (Placebo Comparator): Placebo (rice dextrin or similar) taken daily
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Aloe Vera Extract 1 — 2 capsules taken daily for 30 days
  Arms: Manapol
Dietary Supplement: Control — 2 capsules taken daily for 30 days
  Arms: Placebo
Dietary Supplement: Aloe Vera Extract 2 — 2 capsules taken daily for 30 days
  Arms: Dalton Max

SUMMARY:
The present study will compare the effect of Manapol to DaltonMax on select measures of health. Currently, both ingredients are sold both as a stand-alone dietary supplement and as an active ingredient within various multi-nutrient products.

Immune function will be assessed using blood samples to determine white blood cell counts and distributions, and cytokine levels with/without lipopolysaccharide (LPS) challenge. Additionally, effects specific to antioxidant function and glucose regulation, glucose, insulin, lipid peroxidation, and advanced oxidation protein products will be observed. Antioxidant capacity will also be measured. as well as completion of weekly questionnaires regarding gut health, and microbiome analysis.

DETAILED DESCRIPTION:
Previous research has identified many beneficial properties of aloe vera extracts on health including the "induction of apoptosis, hepatoprotection, antioxidant, antibacterial, antidiabetic, antihyperglycemic, and anti-inflammatory effects". Further, aloe vera may ameliorate digestive issues such as irritable bowel syndrome, as indicated in a recent meta-analysis, although findings are somewhat inconsistent across studies and may be dependent on aloe form and dosage.

The present study will compare the effect of Manapol to DaltonMax on select measures of health. Currently, both ingredients are sold both as a stand-alone dietary supplement and as an active ingredient within various multi-nutrient products.

Immune function will be assessed using blood samples to determine white blood cell counts and distributions, and cytokine presence (IL-1β, IL-6, IL-10, TNF-alpha) with/without lipopolysaccharide (LPS) challenge. Additionally, aloe has been noted to have multiple effects specific to antioxidant function and glucose regulation, glucose, insulin, lipid peroxidation, and advanced oxidation protein products. An increase in blood antioxidant capacity was noted in an earlier study of Ambrotose, therefore antioxidant capacity will also be measured. As prior studies of aloe, coupled with anecdotal reports, provide evidence specific to a potential benefit to gut health, subjects will complete weekly questionnaires regarding gut health, and have a microbiome analysis performed.

ELIGIBILITY:
Inclusion Criteria:

* no consumption of alcohol-containing beverages within 48 hours of testing
* no consumption of caffeine-containing beverages within 48 hours of testing
* no strenuous exercise within 48 hours of testing
* be able to fast overnight (>10 hrs)

Exclusion Criteria:

* self-reported active infection or illness of any kind
* diabetic
* diagnosed with an autoimmune disease including but not limited to rheumatoid arthritis, lupus, Multiple sclerosis, Guillain-Barre syndrome, Psoriasis
* diagnosed GI-related health problems
* using tobacco products
* allergic or hypersensitive to aloe vera
* if female, pregnant or lactating
* using antibiotics
* using a medication/dietary supplement that alters immune or digestive function or that might otherwise impact study outcomes including, but not limited to supplements with immune, immunity, or defense in their name, immunosuppressants including Cyclosporines (Neoral®, Gengraf®, Sandimmune®), Tacrolimus (Prograf®, FK506), Mycophenolate mofetil (CellCept®), Prednisone, Azathioprine (Imuran®), Sirolimus (Rapamune®), Daclizumab and Basiliximab (Zenapax® and Simulect®), OKT3® (monoclonal antibody), Anti-Fungal Medications (Mycelex Troche®, Nystatin® Swish and Swallow, and Diflucan®), Antiviral Medications: Zovirax® (acyclovir), Cytovene® (ganciclovir), and Valcyte® (valganciclovir), Diuretics: Lasix® (furosemide), Antibiotics: Bactrim® (septra), Anti-Ulcer Medications: Prilosec® (omeprazole), Prevacid® (lansoprazole), Zantac® (ranitidine), Axid® (nizatidine), Carafate®(sucralfate), Pepcid®

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
White blood cell characterization | baseline
  A blood sample will be used to characterize the white blood cell population (cell count and distribution)
White blood cell characterization | on day 30 of treatment
  A blood sample will be used to characterize the white blood cell population (cell count and distribution)
Cytokine Panel for plasma | baseline
  IL-1beta, IL-6, IL-10, and TNF-alpha will be quantified from plasma
Cytokine Panel for plasma | on day 30 of treatment
  IL-1beta, IL-6, IL-10, and TNF-alpha will be quantified from plasma
Cytokine Panel on LPS stimulated whole blood | baseline
  IL-1beta, IL-6, IL-10, and TNF-alpha will be quantified on whole blood treated with LPS
Cytokine Panel on LPS stimulated whole blood | on day 30 of treatment
  IL-1beta, IL-6, IL-10, and TNF-alpha will be quantified on whole blood treated with LPS
Glucose | baseline
  Glucose levels in blood will be measured
Glucose | on day 30 of treatment
  Glucose levels in blood will be measured
Insulin | baseline
  Insulin levels in a blood sample will be measured
Insulin | on day 30 of treatment
  Insulin levels in a blood sample will be measured
Lipid peroxidation | baseline
  Lipid peroxiation in a blood sample will be quantified
Lipid peroxidation | on day 30 of treatment
  Lipid peroxiation in a blood sample will be quantified
Advanced oxidation protein products | baseline
  Advanced oxidation protein products in a blood sample will be quantified
Advanced oxidation protein products | on day 30 of treatment
  Advanced oxidation protein products in a blood sample will be quantified
Blood antioxidant capacity | baseline
  Blood antioxidant capacity will be quantified from a blood sample
Blood antioxidant capacity | on day 30 of treatment
  Blood antioxidant capacity will be quantified from a blood sample
Self-reported assessment of fatigue & associated variables | baseline
  Subjects will self-report feelings by marking a scale from 0 (None) to 10 (Extreme) for different fatigue associated variables: Attentive, Tired, Alert, Groggy, Focuse, Sluggish, Energetic, Lethargic, Enthusiastic, Sore, Well-rested, Fatigue, Sickly, Mental Stress.
Self-reported assessment of fatigue & associated variables | Week 1 of treatment
  Subjects will self-report feelings by marking a scale from 0 (None) to 10 (Extreme) for different fatigue associated variables: Attentive, Tired, Alert, Groggy, Focuse, Sluggish, Energetic, Lethargic, Enthusiastic, Sore, Well-rested, Fatigue, Sickly, Mental Stress.
Self-reported assessment of fatigue & associated variables | Week 2 of treatment
  Subjects will self-report feelings by marking a scale from 0 (None) to 10 (Extreme) for different fatigue associated variables: Attentive, Tired, Alert, Groggy, Focuse, Sluggish, Energetic, Lethargic, Enthusiastic, Sore, Well-rested, Fatigue, Sickly, Mental Stress.
Self-reported assessment of fatigue & associated variables | Week 3 of treatment
  Subjects will self-report feelings by marking a scale from 0 (None) to 10 (Extreme) for different fatigue associated variables: Attentive, Tired, Alert, Groggy, Focuse, Sluggish, Energetic, Lethargic, Enthusiastic, Sore, Well-rested, Fatigue, Sickly, Mental Stress.
Self-reported assessment of fatigue & associated variables | Week 4 of treatment
  Subjects will self-report feelings by marking a scale from 0 (None) to 10 (Extreme) for different fatigue associated variables: Attentive, Tired, Alert, Groggy, Focuse, Sluggish, Energetic, Lethargic, Enthusiastic, Sore, Well-rested, Fatigue, Sickly, Mental Stress.
Subjects' perceived digestive/bowel health | baseline
  Subjects will record their bowel movements/health using the Bristol stool chart weekly and questionnaire on their upper abdominal, lower abdominal, and other digestive symptoms on a scale 0 (no problem at all) to 9 (the worst it has ever been)
Subjects' perceived digestive/bowel health | Week 1 of treatment
  Subjects will record their bowel movements/health using the Bristol stool chart weekly and questionnaire on their upper abdominal, lower abdominal, and other digestive symptoms on a scale 0 (no problem at all) to 9 (the worst it has ever been)
Subjects' perceived digestive/bowel health | Week 2 of treatment
  Subjects will record their bowel movements/health using the Bristol stool chart weekly and questionnaire on their upper abdominal, lower abdominal, and other digestive symptoms on a scale 0 (no problem at all) to 9 (the worst it has ever been)
Subjects' perceived digestive/bowel health | Week 3 of treatment
  Subjects will record their bowel movements/health using the Bristol stool chart weekly and questionnaire on their upper abdominal, lower abdominal, and other digestive symptoms on a scale 0 (no problem at all) to 9 (the worst it has ever been)
Subjects' perceived digestive/bowel health | Week 4 of treatment
  Subjects will record their bowel movements/health using the Bristol stool chart weekly and questionnaire on their upper abdominal, lower abdominal, and other digestive symptoms on a scale 0 (no problem at all) to 9 (the worst it has ever been)
Microbiome analysis | baseline
  Subjects will submit a stool sample kit for microbiome analysis
Microbiome analysis | on Day 30 of treatment
  Subjects will submit a stool sample kit for microbiome analysis

SECONDARY OUTCOMES:
Food Logs | baseline
  Subjects will record their dietary consumption for the 5 days leading up to each test visit
Food Logs | on Day 30 of treatment
  Subjects will record their dietary consumption for the 5 days leading up to each test visit
Resting Blood Pressure | baseline
  Blood pressure will be measured following a 10 min rest using an automated system
Resting Blood Pressure | on Day 30 of treatment
  Blood pressure will be measured following a 10 min rest using an automated system
Resting Heart Rate | baseline
  Heart rate will be measured following a 10 min rest using an automated system
Resting Heart Rate | on day 30 of treatment
  Heart rate will be measured following a 10 min rest using an automated system

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bloomer, PhD, Principal Investigator — University of Memphis
Locations (1):
- Center for Nutraceutical and Dietary Supplement Research, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No